CLINICAL TRIAL: NCT04086160
Title: Effects of Transcranial Direct Current Stimulation (tDCS) on Motor Function in Schizophrenia Patients and Individuals at Risk for Psychotic Onset
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr WANG Shumei (Other)
Responsible Party: Sponsor-Investigator, Dr WANG Shumei, Assistant Professor, The Hong Kong Polytechnic University
Organization: The Hong Kong Polytechnic University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20190518001
Record Dates: First submitted 2019-07-27; First posted 2019-09-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia; Psychosis; Parkinsonism; Dyskinesias
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Parkinsonian Disorders; Dyskinesias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- schizophrenia- tDCS (Experimental)
  Interventions: Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY)
- schizophrenia- sham (Sham Comparator)
  Interventions: Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY)
- at risk- tDCS (Experimental)
  Interventions: Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY)
- at risk- sham (Sham Comparator)
  Interventions: Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY)
- healthy controls for schizophrenia- tDCS (Experimental)
  Interventions: Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY)
- healthy controls for schizophrenia- sham (Sham Comparator)
  Interventions: Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY)
- healthy controls for at risk- tDCS (Experimental)
  Interventions: Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY)
- healthy controls for at risk- sham (Sham Comparator)
  Interventions: Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY)

INTERVENTIONS:
Device: Transcranial direct current stimulation device (Soterix Medical, New York, NY) — Transcranial direct current stimulation (tDCS) is a non-invasive intervention, which applies low-amplitude direct electric currents to the brain through scalp electrodes. The real (2mA) or sham tDCS intervention will be given for a total of eight sessions in four weeks with 20 minutes per session.

SUMMARY:
The purposes of this research are to investigate (1) if schizophrenia patients and at-risk individuals present bradykinesia and dyskinesia and (2) if tDCS improves motor performance in schizophrenia patients and at-risk individuals. The first hypothesis is that both schizophrenia patients and at-risk individuals show bradykinesia and dyskinesia, and the motor symptoms are more severe in the former than the latter. The second hypothesis is that tDCS improves motor performance in schizophrenia patients and at-risk cases.

ELIGIBILITY:
Inclusion Criteria for schizophrenia patients:

* a diagnosis of schizophrenia without other psychiatric diseases
* having stable psychotic symptoms
* a score of 22 or above in Hong Kong version Montreal Cognitive Assessment
* having no neurological diseases and no medical conditions that affect motor performance

No Exclusion Criteria.

Inclusion Criteria for at-risk individuals:

* a score of nine or above in the Chinese version of the 16-item Prodromal Questionnaire (CPQ-16)
* a score of 22 or above in Hong Kong version Montreal Cognitive Assessment
* having no diagnosis of psychiatric diseases
* having no neurological diseases and no medical conditions that affect motor performance

No Exclusion Criteria.

Inclusion Criteria for healthy controls:

* a score less than nine in CPQ-16
* a score of 22 or above in Hong Kong version Montreal Cognitive Assessment
* having no diagnosis of psychiatric diseases
* having no neurological diseases and no medical conditions that affect motor performance.

No Exclusion Criteria.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right before the 1st session of tDCS
  normalized movement time (representing severity of parkinsonism). Unit: second/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right after the 8th (last) session of tDCS
  normalized movement time (representing severity of parkinsonism). Unit: second/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right before the 1st session of tDCS
  normalized number of movement units (representing severity of dyskinesia). Unit: units/mm
Motion analysis by using an eight-camera motion capture system (VICON; Oxford Metrics Group, Oxford, UK) | Within one week right after the 8th (last) session of tDCS
  normalized number of movement units (representing severity of dyskinesia). Unit: units/mm

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No